CLINICAL TRIAL: NCT06651775
Title: Effectiveness of High Intensity Laser Therapy (HILT) in Patients With Chronic Lumbar Radiculopathy Due to Disc Herniation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Talha Yılmaz, medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2-24-6770
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Radiculopathy
Keywords: Activity of Daily Living; chronic low back pain; high intensity laser therapy; pain
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT group (Experimental): Receiving Hotpack+TENS+Exercises+HILT
  Interventions: Device: High intensity laser therapy
- Sham group (Sham Comparator): Receiving Hotpack+TENS+Exercises+ sham HILT
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: High intensity laser therapy — lumbosciatalgia mode of the HILT device
  Arms: HILT group
Device: Sham Comparator — sham mode of the HILT device
  Arms: Sham group

SUMMARY:
The aim of the researchers in this intervention study was to see the effects of High Intensity Laser Therapy (HILT) on participants' disability, functionality and pain parameters in chronic radicular low back pain due to lumbar disc herniation, and to investigate its superiority over widely used conventional electrotherapy modalities.

The main question it aims to answer is:

What is the short and long term effect of high intensity laser therapy on low back and leg pain in patients with chronic lumbar radiculopathy due to disc herniation?

35 patients in group A will receive the planned Hotpack, TENS, High Intensity Laser Therapy (HILT) and exercise treatments for lumbar radicular low back pain. In group B (comparison group) 35 patients will receive Hotpack, TENS, sham HILT, and exercise treatments.

Participants will receive 15 sessions of treatment and exercises will be given as a home program. Both groups will complete questionnaires about disability, life functions and pain before and after treatment and at the 3rd month follow-up.

DETAILED DESCRIPTION:
Efficacy of High Intensity Laser Therapy in Patients with Chronic Lumbar Radiculopathy Due to Disc Herniation , Ankara 2025

Low back pain is an important and widespread health problem that negatively affects the quality of life from past to present, causes deterioration in functional status and may cause disability and psychologically wears out human health in the chronic period. In epidemiological studies, the prevalence of low back pain has been found to be approximately 40% throughout life.

Low back pain is classified as acute, subacute and chronic according to its duration and as mechanical and inflammatory according to the character of the pain. Low back pain lasting more than 12 weeks is defined as chronic low back pain.

Etiological factors include fracture, malignancy, infection, trauma, osteoporosis, inflammatory diseases, myogenic causes, etc. One of the most important and common causes of mechanical causes is intervertebral disc herniation. Disc herniation may also cause radicular pain in the form of numbness, burning, electrification, pins and needles in the dermatome area of the related nerve due to neural root compression.

There are many treatment modalities for radicular low back pain due to lumbar disc herniation. These include medical treatment, lumbar and abdominal strengthening exercises given outside the acute painful period, physical therapy modalities, alternative medicine methods, laser therapy, epidural steroid injections and surgical treatment.

The term laser is defined as "light amplification by stimulated radiation emission". It is a non-invasive and painless treatment. There are two types of laser therapy, low and high intensity, with different intensity according to peak power and wavelength. Pulsed neodymium-doped yttrium aluminium garnet (Nd:YAG) high intensity laser, HILT, works with high peak power and 1.064nm wavelength. The laser has 5 basic mechanisms of action: thermal, mechanical, electrical, photochemical, biostimulate. Biostimulation, antiedema, analgesic and anti-inflammatory effects in the applied area are more pronounced due to its high intensity and specific wavelength, but the exact mechanism of action in reducing pain has not yet been clearly clarified.

This study, aimed to investigate the effects of high-intensity laser therapy (HILT) on the patient's disability, functionality, and neuropathic and nociceptive patterns of pain in radicular pain due to lumbar disc herniation in the chronic period and its superiority over the conventional electrotherapy modalities we frequently use. The study was designed as a randomised, placebo-controlled, double-blind, prospective study.

This study includes patients admitted to the outpatient clinics of Ankara City Hospital Physical Medicine and Rehabilitation Hospital who have low back pain radiating to the lower extremities for more than 12 weeks and have sensory deficit and/or pain sensation in dermatomal distribution due to radicular lesion accompanying lumbar disc herniation shown by lumbar MRI. Patients will be randomly divided into two groups.

A total of 70 patients aged 18-65 years of male and female sex will be included in the study and the patients will be randomly divided into two groups of equal number.

Patients in Group A (n:35) will receive 15 sessions of hotpack and 15 sessions of TENS (transcutaneous electrical nerve stimulation) five days a week for 3 weeks, 15 sessions of HIRO TT (ASA Laser, Arcugnano, Italy) device in lumbosciatica mode in three phases (fast scanning, trigger point, slow scanning) over an area of 25 cm². Isometric lumbar strengthening and core stabilisation exercises will be given to the patients as a home programme.

Patients in group B (n:35) will receive TENS (Transcutaneous Electrical Nerve Stimulation), Hotpack, Lumbar and Core Stabilisation Exercises and sham High Intensity Laser treatments and the protocols will be the same as in group A. Patients will be evaluated 3 times in total: pre-treatment, post-treatment and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lumbar radiculopathy due to lumbar disc herniation and whose complaints are correlated with lumbar MRI
* Patients aged 18-65 years
* Patients who agreed to participate in the study
* Literate patients

Exclusion Criteria:

* Pregnancy
* Patients with cardiac pacemakers
* Patients with a diagnosis of inflammatory rheumatic disease,
* Patients with a diagnosis of polyneuropathy that precludes receiving treatment,
* Patients with active or history of malignancy within the last 1 year and currently receiving chemotherapy and/or radiotherapy,
* Patients with serious psychiatric illness,
* Patients with severe coagulation disorders,
* Spinal Stenosis (patients with spinal canal diameter less than 8 mm)
* Patients with neurologic deficits that prevent them from receiving treatment,
* Patients with active infection,
* Patients with vasculitis,
* Patients with skin disease in the treated area,
* Patients who received steroid injections and/or physical therapy for the lumbar region within the last 3 months,
* Patients undergoing lumbar spine surgery,
* Patients with acute trauma,
* Patients with a history of lumbar instability,
* Patients with uncontrolled or severe cardiovascular or metabolic disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | pre-treatment, immediately post-treatment and three months follow-up
  Visual Analogue Scale (VAS) is used to convert some values that cannot be measured numerically into numerical form. On the two ends of a 100 mm line, two extreme definitions of the parameter to be evaluated are written and the patient is asked to indicate where his/her condition is appropriate on this line by drawing a line or putting a point or pointing. For example, for pain, no pain is written on one end, very severe pain is written on the other end and the patient marks his/her current situation on this line. The length of the distance from the point of no pain to the point marked by the patient indicates the patient's pain. The test has proven itself for a very long time and is recognised in the world literature. In our study, the VAS values of the patients for low back and leg pain at rest and in motion will be questioned and followed up.
Revised Oswestry Disability Index (ODI) | pre-treatment, immediately post-treatment and three months follow-up
  It was developed to assess the degree of loss of function in low back pain. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleeping, the degree of change in pain, travelling and social life. Under each item, there are six statements that the patient marks the appropriate one for his/her condition. The first statement is scored as "0" and the sixth statement as "5". When the total score is calculated, it is multiplied by two and expressed as a percentage. The maximum score is "100" and the minimum score is "0". The higher the total score, the higher the level of disability. Revised Oswestry Disability Index (ODI) consists of 10 items. Turkish validity and reliability was demonstrated in 2004.

SECONDARY OUTCOMES:
Nottingham Health Profile (NHP) | pre-treatment, immediately post-treatment and three months follow-up
  This questionnaire includes 38 items assessing quality of life in 6 sections (pain, energy level, sleep, social isolation, emotional reaction, physical activity). Physical mobility (8 questions), pain (8 questions), sleep (5 questions), emotional reactions (9 questions), social isolation (5 questions) The evaluation was made by taking the percentage of yes answers. Each section is scored between 0 and 100. 0 indicates the best score and 100 indicates the worst score. Turkish validation of the NHP was conducted by Kucukdeveci AA. et al.
LANSS Pain Scale | pre-treatment, immediately post-treatment and three months follow-up
  The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale is a scale based on the analysis of data obtained during bedside examination. First used by Bennett, the LANSS Pain Scale is a very useful tool that provides immediate information in the clinical setting and helps to differentiate nociceptive pain from neuropathic pain. The LANSS Pain Scale is categorised in the range of 0-24 points. A score of 12 or more is in favour of neuropathic pain and a score below 12 is in favour of nociceptive pain. Turkish validity and reliability have been proven.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
only study protocol
Supporting Information: Study Protocol